CLINICAL TRIAL: NCT07005102
Title: A Phase 2/3 Randomized Study to Evaluate the Safety, Efficacy, and Optimal Dose of Telisotuzumab Adizutecan in Combination With Osimertinib as First-Line Treatment in Patients With Locally Advanced Unresectable or Metastatic EGFR-Mutated Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study to Assess Adverse Events, Change in Disease Activity of Intravenous Telisotuzumab Adizutecan in Combination With Osimertinib as First-Line Treatment in Adult Participants With Locally Advanced Unresectable or Metastatic EGFR-Mutated Non-Squamous Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M25-287; 2024-518586-10 (Other: EU CT)
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
Keywords: Non-Squamous Non-Small Cell Lung Cancer; Telisotuzumab Adizutecan; Osimertinib; ABBV-400, Stand of Care; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care; osimertinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Stage 1: Escalation Telisotuzumab Adizutecan with Osimertinib (Experimental): Participants will receive increasing doses of telisotuzumab adizutecan with osimertinib (Osi), as part of the approximately 76 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Osimertinib (Osi)
- Stage 1: Expansion Telisotuzumab Adizutecan Dose A with Osi (Experimental): Participants will receive telisotuzumab adizutecan dose A with Osi, as part of the approximately 76 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Osimertinib (Osi)
- Stage 1: Expansion Telisotuzumab Adizutecan Dose B with Osi (Experimental): Participants will receive telisotuzumab adizutecan dose B with Osi, as part of the approximately 76 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Osimertinib (Osi)
- Stage 1: Expansion Telisotuzumab Adizutecan Dose C with Osi (Experimental): Participants will receive telisotuzumab adizutecan dose C with Osi, as part of the approximately 76 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Osimertinib (Osi)
- Stage 1: Expansion Osi (Experimental): Participants will receive Osi, as part of the approximately 76 month study duration.
  Interventions: Drug: Osimertinib (Osi)
- Stage 2: Standared of Care (SOC) Osi (Experimental): Participants will receive Osi, as part of the approximately 76 month study duration.
  Interventions: Drug: Standard of Care
- Stage 2: Telisotuzumab Adizutecan Optimized with Osi (Experimental): Participants will receive the optimized dose of telisotuzumab adizutecan with Osi, as part of the approximately 76 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Osimertinib (Osi)

INTERVENTIONS:
Drug: Standard of Care — Standard of Care
  Arms: Stage 2: Standared of Care (SOC) Osi
Drug: Telisotuzumab Adizutecan — Intravenous (IV) Infusion
  Arms: Stage 1: Escalation Telisotuzumab Adizutecan with Osimertinib; Stage 1: Expansion Telisotuzumab Adizutecan Dose A with Osi; Stage 1: Expansion Telisotuzumab Adizutecan Dose B with Osi; Stage 1: Expansion Telisotuzumab Adizutecan Dose C with Osi; Stage 2: Telisotuzumab Adizutecan Optimized with Osi
Drug: Osimertinib (Osi) — Oral Tablet
  Arms: Stage 1: Escalation Telisotuzumab Adizutecan with Osimertinib; Stage 1: Expansion Osi; Stage 1: Expansion Telisotuzumab Adizutecan Dose A with Osi; Stage 1: Expansion Telisotuzumab Adizutecan Dose B with Osi; Stage 1: Expansion Telisotuzumab Adizutecan Dose C with Osi; Stage 2: Telisotuzumab Adizutecan Optimized with Osi

SUMMARY:
Non-small cell lung cancer (NSCLC) is a common type of lung cancer where abnormal cells in the lungs grow out of control. The purpose of this study is to assess adverse events and change in disease activity when telisotuzumab adizutecan is given in combination with a fixed dose of osimertinib (Osi), Osi alone, or standard of care (SOC) alone.

Telisotuzumab adizutecan is an investigational drug being developed for the treatment of NSCLC. Osi is a drug approved for the treatment of NSCLC. This study will be divided into two stages, in the first stage participants will receive increasing doses of telisotuzumab adizutecan with Osi. Participants will then be randomized into 4 groups called treatment arms where 3 groups will receive 1 of 3 optimized doses of telisotuzumab adizutecan from the dose escalation phase with Osi, or Osi alone. In the second stage participants will receive the optimal dose of telisotuzumab adizutecan, from the previous stage, with Osi, or SOC. Approximately 694 adult participants with mCRC will be enrolled in the study in 200 sites worldwide.

In Stage 1, during dose escalation participants will receive increasing intravenous (IV) doses of telisotuzumab adizutecan with oral Osi tablets. During dose optimization participants will receive OSi alone or with 1 of 3 optimized doses of telisotuzumab adizutecan. In stage 2 participnats will recieve the optimal dose of IV telisotuzumab adizutecanin with oral Osi tablet, or SOC. The study will run for a duration of approximately 76 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 during the screening period and prior to dosing of study treatment on Cycle 1 Day 1.
* Must consent to provide recently obtained formalin-fixed, paraffin-embedded (FFPE) tumor tissue (ideally collected during or after locally advanced or metastatic diagnosis) or archived tissue during screening for c-Met immunohistochemistry (IHC) testing and study stratification. c-Met IHC results are required prior to randomization.
* Must have at least one non-irradiated measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. If only one measurable lesion exists, it is acceptable to be used (as a target lesion) as long as it has not been previously irradiated and as long as it has not been biopsied within 14 days of the baseline tumor assessment scans.
* Any toxicities from prior systemic anti-cancer therapy must have resolved to common terminology criteria for adverse events (CTCAE) Grade 1 or baseline level (except for alopecia [any grade] or Grade <= 2 peripheral neuropathy).
* Should not have any major, life-threatening conditions and life expectancy as determined by the investigator should be at least 3 months.

Exclusion Criteria:

* History of interstitial lung disease (ILD), pneumonitis that required treatment with systemic steroids, or any evidence of active ILD/pneumonitis on screening chest computed tomography (CT) scan.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis.
* Participants has leptomeningeal disease, or subject has spinal cord compression not definitively treated with surgery or radiation.
* History of any malignancy except for malignancy treated with curative intent and with no known active disease present for 2 years before the first dose of study treatment and felt to be at low risk for recurrence by investigator, successfully treated nonmelanoma skin cancer or localized carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 694 (Estimated)
Dates: Start 2025-08-03 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Objective Response (OR) Based on Blinded Independent Central Review (BICR) Assessment per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to Approximately 76 Months
  OR is defined as confirmed complete response (CR) or confirmed partial response (PR) per BICR based on RECIST version 1.1.
Phase 3: Progression-free survival (PFS) based on BICR assessment per RECIST version 1.1. | Up to Approximately 76 Months
  PFS is defined as the time from the participant's randomization date to the first occurrence of radiographic progression per BICR based on RECIST version 1.1 or death from any cause, whichever occurs earlier.
Number of Participants with Adverse Events (AEs) | Up to Approximately 76 Months
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Phase 2: PFS based on BICR assessment per RECIST version 1.1. | Up to Approximately 76 Months
  PFS is defined as the time from the participant's randomization date to the first occurrence of radiographic progression per BICR based on RECIST version 1.1 or death from any cause, whichever occurs earlier.
Phase 2: Duration of response (DoR) based on BICR assessment per RECIST version 1.1. | Up to Approximately 76 Months
  DOR is defined as the time from the first documented CR or PR per BICR to the first occurrence of radiographic progression per RECIST version 1.1 or death from any cause, whichever occurs first. DOR is defined for participants with confirmed CR/PR.
Phase 2: Disease control rate (DC) based on BICR assessment per RECIST version 1.1. | Up to Approximately 76 Months
  DC is defined as best overall response of confirmed CR or confirmed PR, or stable disease (SD) for at least 12 weeks following randomization date based on RECIST version 1.1, as determined by the BICR.
Phase 2: Overall Survival | Up to Approximately 76 Months
  OS is defined as the time from participant's randomization date to the event of death from any cause.
Phase 3: Overall Survival | Up to Approximately 76 Months
  OS is defined as the time from participant's randomization date to the event of death from any cause.
Phase 3: OR based on BICR assessment per RECIST version 1.1. | Up to Approximately 76 Months
  OR is defined as confirmed CR or confirmed PR per BICR based on RECIST version 1.1.
Phase 3: DoR based on BICR assessment per RECIST version 1.1. | Up to Approximately 76 Months
  DOR is defined as the time from the first documented CR or PR per BICR to the first occurrence of radiographic progression per RECIST version 1.1 or death from any cause, whichever occurs first. DOR is defined for participants with confirmed CR/PR.
Phase 3: DC based on BICR assessment per RECIST version 1.1. | Up to Approximately 76 Months
  DC is defined as best overall response of confirmed CR or confirmed PR, or SD for at least 12 weeks following randomization date based on RECIST version 1.1, as determined by the BICR.
Phase 3: Change from baseline at Week 12 in physical functioning as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). | Up to Approximately 76 Months
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Phase 3: Change from baseline at Week 12 in key lung cancer symptoms as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 (EORTC QLQ-LC13) | Up to Approximately 76 Months
  The EORTC QLQ-LC13 is a lung cancer specific module and consists of 13 questions assessing lung cancer-associated symptoms and treatment-related effects, including one multiple-item scale to assess dyspnea and a series of single items assessing coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain, and pain medication. Each item is assessed on a Likert scale from 1 (not at all) to 4 (very much).
Phase 3: Change from baseline at Week 12 in GHS/QoL as measured by the EORTC QLQ-C30. | Up to Approximately 76 Months
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (41):
- United States (10):
  - USC Norris Comprehensive Cancer Center /ID# 275343, Los Angeles, California
  - Usc Norris Oncology/Hematology Treatment Center /ID# 278673, Newport Beach, California
  - Mid Florida Hematology And Oncology Center /ID# 275278, Orange City, Florida
  - The Iowa Clinic /ID# 276020, West Des Moines, Iowa
  - Nho - Revive Research Institute /ID# 276115, Lincoln, Nebraska
  - Renown Regional Medical Center /ID# 276049, Reno, Nevada
  - Texas Oncology - South Austin /ID# 276033, Austin, Texas
  - The University of Texas MD Anderson Cancer Center /ID# 275107, Houston, Texas
  - Texas Oncology - Palestine Cancer Center /ID# 276034, Palestine, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 275071, Fairfax, Virginia
- Australia (4):
  - Liverpool Hospital /ID# 276304, Liverpool, New South Wales
  - The Queen Elizabeth Hospital /ID# 275719, Woodville, South Australia
  - Austin Health /ID# 275505, Heidelberg, Victoria
  - St John Of God Murdoch Hospital /ID# 275700, Murdoch, Western Australia
- Belgium (3):
  - Jessa Ziekenhuis - Campus Virga Jesse /ID# 275585, Hasselt, Limburg
  - Universitair Ziekenhuis Leuven /ID# 275586, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 275753, Roeselare, West-Vlaanderen
- Israel (3):
  - The Chaim Sheba Medical Center /ID# 274541, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 274542, Haifa
  - Rabin Medical Center. /ID# 274540, Petah Tikva
- IRCCS Istituti Fisioterapici Ospitalieri-Istituto Nazionale Tumori Regina Elena /ID# 274948, Rome, Roma, Italy
- Japan (4):
  - Yokohama Municipal Citizen's Hospital /ID# 275682, Yokohama, Kanagawa
  - Niigata University Medical & Dental Hospital /ID# 275685, Niigata, Niigata
  - Osaka Medical And Pharmaceutical University Hospital /ID# 275684, Takatsuki, Osaka
  - Juntendo University Hospital /ID# 276424, Bunkyo-ku, Tokyo
- Portugal (3):
  - Unidade Local de Saude de Braga, EPE /ID# 275394, Braga
  - Unidade Local de Saude de Santo Antonio, E.P.E. /ID# 275387, Porto
  - Hospital Cuf Porto /ID# 275395, Porto
- Singapore (2):
  - National Cancer Centre Singapore /ID# 275986, Singapore, Central Singapore
  - National University Hospital /ID# 275988, Singapore
- South Korea (5):
  - Inje University Haeundae Paik Hospital /ID# 275388, Busan, Busan Gwang Yeogsi
  - Chungbuk National University Hospital /ID# 275768, Cheongju-si, North Chungcheong
  - Yonsei University Health System Severance Hospital /ID# 275384, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 275600, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 278083, Seoul, Seoul Teugbyeolsi
- Spain (3):
  - Hospital Clinic de Barcelona /ID# 275476, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 275475, Madrid
  - Instituto Valenciano de Oncología /ID# 275471, Valencia
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 275293, Kaohsiung City
  - National Taiwan University Cancer Center (Ntucc) /ID# 275291, Taipei
  - Taipei Veterans General Hospital /ID# 275292, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-311